CLINICAL TRIAL: NCT01576471
Title: A Phase II Study to Evaluate the Efficacy and Safety of 12 Weeks of Treatment With Oral CNDO 201 Trichuris Suis Ova Suspension (TSO) as Compared to Placebo, Followed by a 12 Week Open-label Treatment Period in Patients With Moderately to Severely Active Crohn's Disease
Brief Title: Efficacy and Safety of Trichuris Suis Ova (TSO) as Compared to Placebo
Acronym: TRUST-I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Coronado Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNDO 201-003
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-04

CONDITIONS: Crohn's Disease
Keywords: T. suis ova; Trichuris suis ova; Inflammatory Bowel Disease; TRUST-I; TRUSTI; TRUST-1; TRUST1
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- TSO 7500 (Experimental)
  Interventions: Biological: Trichuris suis ova (TSO)

INTERVENTIONS:
Biological: Trichuris suis ova (TSO) — TSO 7500: 7500 embryonated, viable TSO every 2 weeks X 10 weeks (up to 6 total doses)
  Arms: TSO 7500
Biological: Placebo — Placebo: dose every 2 weeks X 10 weeks (up to 6 total doses)
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter, and proof of concept study with a parallel group design to evaluate the safety and efficacy of oral Trichuris Suis Ova (TSO) suspension, as compared to placebo, in patients with moderately to severely active Crohn's disease. This study will also have an optional open-label extension for patients completing the double-blind phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female, 18 to 65 years old.
2. Patient with established diagnosis of Crohn's disease (CD) for at least 3 months confirmed by endoscopic and histological, or endoscopic and radiological criteria.
3. Patient with localization of CD either in terminal ileum (L1), in colon (L2) or ileocolitis (L3), all without upper gastrointestinal involvement (- L4) according to the Montreal classification (2005).
4. Patient with active, symptomatic CD manifested by CDAI ≥ 220 and ≤ 450 at Baseline.
5. Patient with active intestinal inflammation as visualized by endoscopy within 8 weeks prior to Baseline.
6. Patient is not using concomitant medication for treatment of underlying Crohn's disease with the following exceptions: concomitant medications may include: 1) Oral or rectal sulfasalazine, mesalazine (5-ASA), or mesalazine derivative, if receiving it for >6 weeks and if receiving the same dose for at least 4 weeks; 2) Oral prednisone up to 15 mg/day, or budesonide if receiving it for >4 weeks and if receiving the same dose for at least 4 weeks; and 3) Azathioprine (up to 2.5 mg/kg daily) or 6-mercaptopurine (up to 2 mg/kg daily) if receiving it for >3 months and if receiving the same dose for at least 8 weeks prior to Baseline.
7. Hemoglobin of at least 10 g/dl, normal white blood cell and platelet count > lower limit of normal at screening.
8. For females of childbearing potential, negative serum pregnancy test prior to enrollment, not breastfeeding for study duration, and willingness to use accepted forms of reliable birth control for study duration [including bilateral tubal ligation, use of oral contraceptives, double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam), Depo-Provera®, hormonal implants, and total abstinence]. Pregnancy tests are not required (indicate "N/A") for males or females not of childbearing potential (post-menopausal with last menstrual period >1 year ago or total hysterectomy).
9. Patient has the ability to provide informed consent.

Exclusion Criteria:

1. Patient with known Crohn's lesions in the upper GI-tract (esophagus, stomach, duodenum, jejunum) with present symptoms.
2. Patient with ulcerative colitis, indeterminate colitis, or ulcerative proctitis.
3. Bowel surgery in past 6 months prior to Screening.
4. Resection of more than 50 cm of the ileum.
5. Current ileostomy or colostomy.
6. Ongoing or active septic complications, is hospitalized or exhibiting signs of toxicity (sepsis), has symptomatic strictures, or impending obstruction or anticipating a need for blood transfusion for gastrointestinal bleeding or in whom surgical intervention may be imminent.
7. Patient with gastrointestinal abscess or perforation.
8. Patient with fistulae having a new onset within 2 months of Screening with moderate to severe local inflammation.
9. Patient with history of colorectal cancer or colorectal dysplasia. Patients with completely resected sporadic adenomas may be enrolled.
10. Patient requiring parenteral or tube feeding.
11. Patient with current evidence of infectious colitis, e.g., Clostridium difficile, Amoebiasis, Giardia lamblia or stools positive for other enteric pathogens, ova or parasites at Screening.
12. Female patient who is pregnant or breastfeeding or wishing to become pregnant during study participation or unwilling to use birth control.
13. Patient with serum creatinine ≥ 2.0 mg/dL; blood urea nitrogen >40 mg/dL; alkaline phosphatase > 250 U/L; aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 100 U/L; or total bilirubin >1.5 mg/dL.
14. Patient with hepatitis B virus, hepatitis C virus, liver cirrhosis or portal hypertension, or is known to be human immunodeficiency virus (HIV) positive.
15. Patient with primary sclerosing cholangitis.
16. Patient with malignancy within the past 5 years, with the exception of completely excised squamous or basal cell skin cancers, and cervical carcinoma in situ.
17. Patient received cyclosporine, an anti-TNFα or other immunomodulatory agents other than azathioprine/6-mercaptopurine within 12 weeks prior to Screening.
18. Patient is a primary non-responder an anti-TNFα.
19. Patient is refractory to azathioprine/6-mercaptopurine.
20. Patient received methotrexate within 6 weeks prior to Screening.
21. Patient received metronidazole within 2 weeks prior to Screening.
22. Patient received non-steroidal anti-inflammatory drugs (NSAIDS) within 2 weeks before Baseline visit for more than 3 consecutive days, except acetylsalicylic acid ≤ 350 mg/d which is allowed.
23. Patient received antibiotic, antifungal or antiparasitic medication in the last 2 weeks prior to Screening and/or would potentially require this during the study treatment period.
24. Patient with history of drug or alcohol abuse within 6 months prior to Screening.
25. Patient with evidence of poor compliance with medical advice and instruction including diet or medication.
26. Patient is unable or unwilling to swallow study medication suspension.
27. Patient with a significant medical condition which puts the patient at risk for study participation and/or for any reason is considered by the Investigator to be an unsuitable patient to receive CNDO-201 TSO or is potentially put at risk by study procedures.
28. Patient who has participated in another clinical trial within 30 days of Screening for this trial and/or any experimental treatment for this population.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nova Silver, Study Director — Coronado Biosciences
Locations (73):
- United States (73):
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - Lynn Institue of the Ozarks, Little Rock, Arkansas
  - Preferred Research Partners, Little Rock, Arkansas
  - Anaheim Clinical Trials, Anaheim, California
  - Rokay Kamyar, MD Inc, La Mesa, California
  - Medvin Clinical Research, La Mirada, California
  - Lakewood Primary Care Medical Group, Inc, Lakewood, California
  - Alliance Research, Long Beach, California
  - Collaborative Neuroscience Network, Inc., Long Beach, California
  - Alliance Clinical Research, LLC, Oceanside, California
  - Digestive Care Associates, San Carlos, California
  - San Diego Clinical Trials, San Diego, California
  - Gastroenterology of the Rockies, Lafayette, Colorado
  - Clinical Research of West Florida, Clearwater, Florida
  - Sanitas Research, Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Florida Medical Research Institute, Gainesville, Florida
  - The Center for Gastrointestinal Disorders, Hollywood, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Gastroenterology Associates of Osceola, Kissimmee, Florida
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - Paramount Public Health & Research Management Services, Miami, Florida
  - Community Research Foundation, Inc, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Selah Medical Center, Boise, Idaho
  - Northwest Gastroenterologists, Arlington Heights, Illinois
  - Suburban Clinical Research, Bolingbrook, Illinois
  - Suburban Clinical Research, Burr Ridge, Illinois
  - The University of Chicago Hospital, Chicago, Illinois
  - Medisphere Medical Research Center, LLC, Evansville, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cotton O'Neil Digestive Healthcare, Topeka, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health Services, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Beyer Research, Kalamazoo, Michigan
  - Midwest Center for Clinical Research, Lee's Summit, Missouri
  - Center for Digestive and Liver Disease, Mexico, Missouri
  - Billings Clinic Research Center, Billings, Montana
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Reno Clinical Trials, Sparks, Nevada
  - South Jersey Medical Associates, P.A., Blackwood, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Albany Medical Center, Albany, New York
  - Digestive Health Physicians, Cheektowaga, New York
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Metropolitan Research Associates, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Clinical Trials of America, Inc., Winston-Salem, North Carolina
  - Consultants for Clinical Research, Inc, Cincinnati, Ohio
  - The Ohio State University-Inflammatory Bowel Disease Ctr, Columbus, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Gastroenterology United of Tulsa, Tulsa, Oklahoma
  - Northwest Gastroenterology Clinic, LLD, Portland, Oregon
  - James J. Boylan Gastroenterology and Liver Diseases, Bethlehem, Pennsylvania
  - Shirish A. Amin, MD, PC, Indiana, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Donald Guthrie Foundation for Education & Research, Sayre, Pennsylvania
  - Cherry Tree Medical, Uniontown, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Austin Gastroenterology PA/Professional Quality Research, Inc, Austin, Texas
  - Lovelace Scientific Resources, Inc., Austin, Texas
  - Diagnostic Clinic of Houston, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Gastroenterology Associates of Northern Virginia, Fairfax, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Wenatchee Valley Medical Center, Wenatchee, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | TSO 7500
Started | 125 | 125
Completed | 117 | 116
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TSO 7500 | Total
Number analyzed (Participants) | 125 | 125 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 125 | 125 | 250
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (1.07) | 40.9 (1.04) | 39.8 (0.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 71 | 132
  Male | 64 | 54 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 13 | 28
  Not Hispanic or Latino | 110 | 112 | 222
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 112 | 117 | 229
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 125 | 125 | 250

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Effects of TSO on the Induction of Response in Crohn's Disease, as Measured Primarily by Crohn's Disease Activity Index (CDAI)
Description: CDAI >= 100 point reduction from baseline
Time Frame: 12 weeks
Population: all patients randomized and treated with at least 1 dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TSO 7500
Number analyzed (Participants) | 125 | 125
Participants | 55 | 58

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: no difference
Arm/Group | Placebo | TSO 7500
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/125
Serious Adverse Events (participants affected / at risk) | 6/125 | 3/125
Other Adverse Events (participants affected / at risk) | 27/125 | 31/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=125) | TSO 7500 (N=125)
Food Poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's Disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abscess Intestinal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Vein disorder (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=125) | TSO 7500 (N=125)
Nausea (Gastrointestinal disorders) | 7 (7) | 10 (10)
Abdominal Pain (Gastrointestinal disorders) | 14 (14) | 14 (14)
Crohn's Disease (Gastrointestinal disorders) | 6 (6) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As specified in each clinical trial agreement